CLINICAL TRIAL: NCT05160831
Title: Human Umbilical Cord Mesenchymal Stem Cells in the Treatment of Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Liu Yang, MD, Professor of Center for Joint Surgery, Southwest Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCforKneeOA
Record Dates: First submitted 2021-12-06; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Knee Osteoarthritis
Keywords: knee joint; osteoarthritis; human umbilical cord mesenchymal stem cells
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human umbilical cord mesenchymal stem cells (Experimental): Human umbilical cord mesenchymal stem cells injection is applied for knee OA patients.
  Interventions: Biological: Human umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: Human umbilical cord mesenchymal stem cells — Human umbilical cord mesenchymal stem cell injection is applied for treating knee OA patients.

SUMMARY:
This study aims to investigate the effectiveness and safety of human umbilical cord mesenchymal stem cell injection in the articular cavity to treat moderate to severe knee osteoarthritis (OA), and whether it can achieve articular cartilage regeneration, reduction of joint pain, and restoration of joint function.

DETAILED DESCRIPTION:
There are more than 100 types of arthritis, and the most common ones are rheumatoid arthritis (RA) and osteoarthritis (OA). The main cause of its pathogenesis is the compensatory hyperplasia of the articular cartilage caused by the body's degenerative changes, which will eventually cause the joint to partially or completely lose its function.

In the past few decades, continuous efforts have been made to treat OA. The treatment of OA changes with the development of the patient's condition. At present, there are many diagnosis and treatment options for knee OA, including conservative treatment and surgical treatment. There is an urgent need for an effective treatment to postpone or terminate the course of OA.

Cell therapy for OA has developed rapidly in recent years and has received widespread attention. Mesenchymal stem cells (MSCs) are pluripotent stem cells with potential of self-renewal, proliferation and differentiation. Stem cells are extracted from the patient's body and then implanted back. Their ability of regeneration and reproduction can fill the damaged cartilage tissue, so as to achieve an effective treatment of the joint damage.

This study aims to investigate the effectiveness and safety of human umbilical cord mesenchymal stem cell injection in the articular cavity to treat moderate to severe knee osteoarthritis (OA), and whether it can achieve articular cartilage regeneration, reduction of joint pain, and restoration of joint function.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have no major organ dysfunction.
* Diagnosed as moderate to severe knee osteoarthritis according to internationally recognized criteria: a). Meets the criteria of the "Guidelines for the Diagnosis and Treatment of Osteoarthritis (2018 Edition)" revised by the Chinese Medical Association Rheumatology Branch in 2018; b). Meets the criteria of Grade 3 or more according to the American College of Rheumatology (ACR); c).Meets the criteria of Grade Ⅲ or more according to Kellgren-Lawrence's OA radiology grading standard.
* Those who have the ability to move independently, except those who use wheelchairs, walkers or crutches, and who have no history of mental illness.
* There is no obvious contraindication to articular cavity injection in hematology and biochemical testing.
* No local or systemic infection.
* Subjects and their families understand the clinical trial protocol and agree to participate in the trial, and sign a written Informed Consent.
* Patients whose pain has lasted for more than half a year, and the routine clinical treatment of oral hormones, opioids and other drugs have been ineffective.

Exclusion Criteria:

* Those who are older than 70 years old or younger than 18 years old, or have no full capacity for civil conduct.
* HIV, hepatitis virus or syphilis virus infection or positive serological test.
* Body mass index (BMI) greater than 30 kg/m2.
* Congenital or acquired knee deformity; severe knee arthritis accompanied by severe varus deformity, with varus greater than 10°.
* Pregnant or lactating women, or women of childbearing age who have a positive pregnancy test within 7 days before receiving treatment.
* Complicated with severe cardiovascular and cerebrovascular, liver, kidney, and endocrine, blood system diseases, malignant tumors, allergies, mental disorders, acute infections or local knee joint infections.
* Patients with immunodeficiency.
* Patients with a history of intra-articular injection within 3 months; patients being treated with immunosuppressive agents and glucocorticoids.
* Patients who are still participating in other clinical trials.
* Subjects who refuse to sign Informed Consent or refuse to participate in this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-20 (Estimated); Primary Completion 2023-01-20 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
VAS score | 1, 3, 6, 12 months after injection
  Changes of Visual Analogue Scale (VAS) score after injection

SECONDARY OUTCOMES:
Kellgren-Lawrence score | 1, 3, 6, 12 months after injection
  Changes of Kellgren-Lawrence Score

OTHER OUTCOMES:
Lequesne Index | 1, 3, 6, 12 months after injection
  Changes of the Lequesne Index
WOMAC score | 1, 3, 6, 12 months after injection
  Changes of the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index
Symptom Grading Scale | 1, 3, 6, 12 months after injection
  Changes of Symptom Grading Scale
SF-12 | 1, 3, 6, 12 months after injection
  Changes of the 12-Item Short Form Survey (SF-12)

CONTACTS AND LOCATIONS:
Overall Officials: Liu Yang, MD, Principal Investigator — Center for Joint Surgery, Southwest Hospital, China; Fuyou Wang, MD, Principal Investigator — Center for Joint Surgery, Southwest Hospital, China